CLINICAL TRIAL: NCT01322100
Title: Electrochemotherapy as a Palliative Treatment for Brain Metastases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to slow patient recruitment
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Rigshospitalet, Denmark (Other); Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HJ 1020
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Brain Metastases; CNS Metastases
Keywords: Brain Metastases, CNS Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: The Electroporation System — The Electroporation System comprises of 3 parts: 1.Switch Box, 2. Driver, 3. Brain Probe
Drug: Bleomycin — Bleomycin dosage for i.v. use is 15.000 IU/m2, and is administered 10-30 minutes before the electric pulses. Bleomycin dosage for intratumoral use is either 2.000 IU, 4.000 IU, or 6.000 IU per 3 ml, and 20 % of the calculated tumor volume is injected.

SUMMARY:
Because electrochemotherapy is a quick and effective treatment for cutaneous metastases, a novel electrode device has been developed for treatment in soft tissue such as the brain. Up to 18 patients will be treated in this phase I dose-escalating study of electrochemotherapy for brain metastases. Primary endpoint of the clinical trial is safety and secondary endpoint is efficacy. One brain metastasis is treated once-only with the electrode device guided stereotactically through a burr hole using CT monitoring. The patient will be fully anesthetized during the treatment procedure. Patients are followed up for 6 months with regard to neurological function, Barthel Index, steroid use and adverse effects registration (CTCAE). Tumor response will be evaluated by Magnetic Resonance imaging (MRI).

DETAILED DESCRIPTION:
Electrochemotherapy is a cancer treatment modality comprising of a combination of electrical pulses delivered by electrodes and chemotherapy supplied either intravenously or intratumorally. It is a quick and effective treatment for cutaneous metastases < 3 cm with a complete response rate of 73 % after once-only treatment. The available electrode devices have so far only been applicable for cutaneous tumors. An electrode has now been developed in collaboration with a medico-technical company. An increasing number of cancer patients suffer from metastases to the brain due to e.g. better control of the systemic peripheral cancer disease. The prognosis for patients with brain metastases remains poor and research into new treatments are needed in this field.

Up to 18 patients will be treated in a dose-escalating study of electrochemotherapy for brain metastases. Primary endpoint of the clinical trial is safety and secondary endpoint is efficacy. One brain metastasis is treated once-only with the electrode device guided stereotactically through a burr hole using CT monitoring. The patient will be fully anesthetized during the treatment procedure. Patients are followed up for 6 months with regard to neurological function, Barthel Index, steroid use and adverse effects registration (CTCAE). Tumor response will be evaluated by Magnetic Resonance imaging (MRI).

The first 6 patients will receive an intravenous dose of bleomycin 15.000 IE/m2 before electric pulses. The following patients will receive an additional intratumoral injection of bleomycin of increasing concentration. The electrical pulses will consist of a series of high voltage pulses of 0.1 millisecond duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years.
* Performance status < 2 (ECOG - Eastern Cooperative Oncology Group).
* Diagnosis of brain metastases originated from histological or cytological verified cancer of any histology.
* Patients should have received whole-brain radiation therapy (WBRT) with a time interval of at least 2 months from completion of WBRT until inclusion in this study.
* Patients must have been offered every available standard treatment.
* Brain metastases to be treated must have a diameter of at least 10 millimetres and no more than 27 millimetres.
* Brain metastases to be treated must be accessible for treatment.
* Estimated life expectancy must be more than 3 months.
* Patients must have adequate organ functions:

Adequate bone marrow reserve: Leucocytes (WBC) > 3.0 x 109/l, thrombocytes > 75 x 109/l, hemoglobin > 7 g/dl.

Hepatic: Alkaline phosphate, ALAT or ASAT and bilirubin must not be increased more than 2 times, pp > 40, APTT in normal range. Medical correction is allowed, e.g. correction of low pp using vitamin K.

Renal: if creatinin > 150 micromolar do a GFR examination (Chrome-EDTA).

* Patients must not have a blood pressure (BP) over 180 mm Hg systolic and 110 mm Hg diastolic.
* Sexually active men and women of childbearing potential must use adequate birth control during this study and 6 month after the administration of bleomycin (contraceptive pills, intrauterine devices, injection of prolonged gestagen, subdermal implantation, hormonal vaginal devices, transdermal patches).
* Participating patients must be able to understand the patient information.
* Participating patients must have signed a written informed consent and power of attorney prior to inclusion in this study.

Exclusion Criteria:

* Acute lung infection.
* Previous bleomycin treatment with more than 200.000 IU/m2.
* Previous allergic reaction to bleomycin.
* Allergy towards the sedation used.
* Pregnancy or breastfeeding. Pregnancy in fertile women is excluded by a measurement of HCG in a blood sample. Sterile or infertile women are excluded from the requirement to use anticonception. To be considered sterile or infertile, the patient must have undergone surgical sterilization (vasectomy/bilateral tubectomy, hysterectomy and bilateral ovariectomy) or be post-menopausal defined as the absence of menstruation.
* Treatment with G-CSF (Granulocyte Colony Stimulating Factor) or other cytokines.
* Lung diffusion capacity (DLCO) below normal. DLCO is to be performed in case of suspected (anamnestic or clinical) reduced lung function.
* Physician's assessment that meningeal carcinomatosis (leptomeningeal disease) is a likely cause of the patient's symptoms.
* Treatment with anticoagulants (marevan, marcumar, innohep).
* Allergic to nickel, chrome or cobalt.
* Participation in another clinical study with an experimental drug up to 4 weeks prior to inclusion.
* Illnesses, medical, social or physiological, that may affect the patient's ability to understand the patient information and participate in the follow-up.
* Other serious systemic illnesses (i.e. active infection, abnormal EKG) that the investigator finds may affect the patient's safety and/or ability to complete the study.
* Treatment with Immunosuppressant drugs such as methotrexate and cyclosporine during the study. Treatment with prednisolone is accepted during the study.
* Implanted pacemaker, defibrillators or hearth valve prosthetics.
* Implanted devices such as neurostimulators, eartransplants, insulinpump, metallic tracheostomy.
* Catheters with metal such as Port á cath, Swan Ganz, P-dialysis cath., ventriculoatrial and -peritoneal shunts, bladder cath. with thermo-measurement.
* Metallic clips/prosthetics/magnets from surgery such as neuro- or abdominal clips, tooth- or other prosthetics.
* Disorganised metallic material such as metal fragments in the eyes, shrapnel, gun shot injuries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-04; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety of the trial treatment. This is evaluated by adverse events registrations (CTCAE). | From treatment to last follow up, planned 6 months

SECONDARY OUTCOMES:
Efficacy of the trial treatment. This is evaluated by target tumor response on Magnetic resonance imaging (MRI). | Patients are evaluable 50 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, MD, DMSci, Principal Investigator — Department of Oncology, Herlev Hospital
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev

REFERENCES:
- [Background] Linnert M, Gehl J. Bleomycin treatment of brain tumors: an evaluation. Anticancer Drugs. 2009 Mar;20(3):157-64. doi: 10.1097/CAD.0b013e328325465e. PMID 19396014
- [Background] Gothelf A, Mir LM, Gehl J. Electrochemotherapy: results of cancer treatment using enhanced delivery of bleomycin by electroporation. Cancer Treat Rev. 2003 Oct;29(5):371-87. doi: 10.1016/s0305-7372(03)00073-2. PMID 12972356